CLINICAL TRIAL: NCT06796530
Title: Medium-Chain Acyl-Coa Dehydrogenase Deficiency (MCADD) and Exercise
Brief Title: High Intensity Exercise in Children with MCADD
Acronym: MCADD-EX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0579
Record Dates: First submitted 2025-01-09; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Medium Chain Acyl CoA Dehydrogenase Deficiency
Keywords: MCADD; CPET; high intensity exercise; acylcarnitine
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: One group of MCADD patients and one healthy control group. Both groups undergo the same exercise protocols and metabolic assessments to compare physiological responses and recovery. The MCADD group's responses are compared to those of the control group to analyze differences in metabolic parameters and safety outcomes following high-intensity exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study (Experimental): children aged 8-17 with Medium-Chain Acyl-CoA Dehydrogenase Deficiency (MCADD) or control will undergo CPET and high intensity exercise circuit.
  Interventions: Procedure: Cardiopulmonary exercise test (CPET); Procedure: High-intensity circuit training

INTERVENTIONS:
Procedure: Cardiopulmonary exercise test (CPET) — Participants undergo a CPET on a stationary bike, measuring gas exchange, ECG, and other parameters. The protocol includes 3 minutes of cycling at a constant load (body weight/2 in Watts), followed by a maximal effort test with an incremental load (Ramp protocol body weight (kg) / 4 in Watts per minute).
Procedure: High-intensity circuit training — The patients will undergo a 10-minute warm-up, followed by ~30 high intensity exercise circuit.

SUMMARY:
Medium-chain acyl-CoA dehydrogenase deficiency (MCADD) is a rare genetic disorder affecting the body's ability to break down certain fats (β-oxidation) for energy, leading to symptoms like hypoketotic hypoglycaemia, jaundice, cardiomyopathy and seizures. responsible for the dehydrogenation step of fatty acids with chain lengths between 6 and 12 carbons as they undergo beta-oxidation in the mitochondria. Deficiency in MCAD can result in energy deficiency, the accumulation of acylcarnitine's and low serum carnitine concentrations.

The primary objective of the pilot study is to analyse the effects of high-intensity exercise (cardiopulmonary exercise testing (CPET) & high intensity circuit exercises ) on metabolic parameters and safety. This research is a pilot study comparing four patients with MCADD to four control subjects with the same characteristics. Blood samples are collected for analysis of substrate utilization.

DETAILED DESCRIPTION:
The primary objective of the study is to analyse the effects of high-intensity exercise (CPET & high intensity circuit exercises) on metabolic parameters and safety. Since exercise is tested approximately two hours after a meal, we expect few symptoms, as fat metabolism is only minimally engaged at this intensity. Of interest could be the recovery from exercise, as fat metabolism is presumably activated during this phase.

Each MCADD-patient will attend two experimental visits. On the day of the first visit, the patient will arrive at UZ Gent after 1.5-hours following the meal. After 30 minutes, they will perform a cardiopulmonary exercise test (CPET) on a cycle ergometer. The standard CPET protocol that will be used is as follows: first, three minutes of cycling at a constant load (body weight (kg) / 2) in Watts), followed by a maximal exercise test (Ramp protocol: (body weight (kg) / 4) in Watts per minute). During the cycling test, gas exchange (spirometry) is measured, and an ECG is taken. If no symptoms are observed, the patient may return home. On the second test day, two hours before the test, a breakfast will be consumed. 1.5-hours following the meal, the patient will arrive at UZ Gent, where a heart monitor will be placed, and an intravenous line will be inserted. Following this, the patient will undergo a high-intensity exercise circuit. Blood samples will be taken before and after the exercise at various intervals: immediately, after 30 minutes, 1 hour, and 1.5-hours. Also, RER will be determined at each timepoint using indirect calorimetry. If no symptoms appear, the patient may return home. The patient will report symptoms for the 48 hours following the test. In the blood samples, measures of substrate utilization will be monitored: Glucose, lactate, acylcarnitine levels, free fatty acids (FFA). Also a marker of muscle damage will be assessed (creatine kinase). Additional measures include: anthropometric measurements, including weight and height, physical activity through the children physical activity questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* 8-17y old
* Control subjects matched by sex, age, and self reported Tanner stage.
* All children: height and weight between P5-P95

Exclusion Criteria:

* No daily medication use
* No conditions other than MCADD that restrict sports participation or physiology (e.g., no heart diseases, diabetes).
* < P5 or > P95 on the height-weight curve
* No neuromotor developmental delay (e.g., delayed achievement of motor milestones)
* No recent immobilization (<6 months)
* No surgeries involving the musculoskeletal system

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
glucose | From start of exercise until 1.5 hours post-exercise.
  Analysis of glucose in blood samples taken before, immediately after, and at intervals (30 minutes, 1 hour, and 1.5 hours) following high-intensity exercise.

SECONDARY OUTCOMES:
Cardiorespiratory response during CPET | During CPET (approximately 30 minutes).
  Measurement of maximal oxygen uptake during the cardiopulmonary exercise test (CPET) on a stationary bike.
Safety: Incidence of adverse events during and after exercise. | During and up to 48 hours post-exercise.
  Monitoring and recording of any symptoms, adverse events, or complications during exercise and the following 48 hours
acylcarnitines | From the end of the exercise circuit until 1.5 hours post-exercise.
  Monitoring of acylcarnitines before and after high intensity exercise

OTHER OUTCOMES:
creatine kinase | From the end of the exercise circuit until 1.5 hours post-exercise.
  Assessment of serum creatine kinase (CK) levels before and after exercise
lactate | From the end of the exercise circuit until 1.5 hours post-exercise.
  Assessment of lactate levels before and after exercise
Fat metabolism during recovery phase. | From the end of the exercise circuit until 1.5 hours post high intensity exercise.
  Monitoring of substrate utilization (including fat metabolism) through measurement of RER.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Verloo, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All anonymous data will be made available upon publication